CLINICAL TRIAL: NCT04284137
Title: Function Improvement Exercises for Older Sedentary Community-dwelling Latino Residents (FE-SaLiR)
Brief Title: FE-SaLiR: Function Improvement Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UTSA#19-250
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Disability Physical; Cognitive Impairment
Keywords: Physical Activity; Qi Gong; Physical Function; Cognitive Function; Mind-body Exercise; Hispanic; Aging Population
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified FE-SaLiR (Experimental): FE-SaLiR is based on modified Ba Duan Jin and Wu Qin Xi exercises that include low to moderate intensity age-tailored activities targeting different parts of the body, integrating breathing and mindfulness. A trained Community Health Worker will serve as the class instructor.
  Interventions: Behavioral: Modified FE-SaLiR
- Unmodified Chinese Medicine Exercise (Experimental): The Ba Duan Jin and Wu Qin Xi low- to moderate- intensity exercises published by the General Administration of Sport of China. A trained Community Health Worker will serve as the class instructor.
  Interventions: Behavioral: Unmodified Chinese Medicine Exercise
- Active Control (Active Comparator): The active control program is a health education program for attention control. The participants will learn knowledge and skills about healthy aging and nutrition in a group with hands-on activities.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Modified FE-SaLiR — Participants will attend a 60-minute exercise program (modified Wu Qin Xi and Ba Duan Jin) in a non-clinical community setting twice a week and will perform the exercises at home using guided video up to three times a week. Text messages will be sent to remind the participants to do the exercise at home.
  Other Names: Modified Group
  Arms: Modified FE-SaLiR
Behavioral: Unmodified Chinese Medicine Exercise — Participants will attend a 60-minute exercise program (Wu Qin Xi and Ba Duan Jin published by the General Administration of Sport of China) in a non-clinical community setting twice a week and will be expected to practice exercise at home using guided video up to three times a week. Text messages will be sent to remind the participants to do the exercise at home.
  Other Names: Unmodified Group
  Arms: Unmodified Chinese Medicine Exercise
Behavioral: Active Control — Participants will attend a 60-minute health education program once a week.
  Other Names: NIH Aging Mastery Program
  Arms: Active Control

SUMMARY:
As complementary and alternative medicines in both Chinese and Western populations, Wu Qin Xi (the Five Animal Play) and Ba Duan Jin (the Eight Pieces of Brocade) have demonstrated small to medium effects on the improvement of various physical, cognitive, and quality of life measures. The purpose of this proposed study is to develop a culturally tailored, low-cost exercise program, "Function Improvement Exercises for Older Sedentary Community-Dwelling Latino Residents (FE-SaLiR)", to improve physical and cognitive functions and quality of life in older Latino adults in a non-clinical community setting. This will be the first study to combine Wu Qin Xi and Ba Duan Jin in non-Chinese population.

The study has three specific aims:

1. Following the community-based participatory research model (CBPR), the research team, community health advocates and senior program participants will co-adapt Wu Qin Xi and Ba Duan Jin and co-design the content and delivery form of FE-SaLiR (Phase 1).
2. To conduct a three-arm pragmatic controlled trial to test the feasibility and acceptability of FE-SaLiR in older sedentary community-dwelling Latino residents (Phase 2).
3. To generate the estimates of effect size and retention from the pilot study data that will be used to conduct the power estimation of a large RCT that will compare the effectiveness of FE-SaLiR with other types of exercises in an NIH RO1 grant application.

FE-SaLiR Phase 1 was delivered from August 2019 to November 2019. FE-SaLiR Phase 2 started recruiting participants by invitation in January 2020; the exercise program started in February 2020.

DETAILED DESCRIPTION:
Phase 1: Formative Study

A 3-month formative study with a community advisory group at the Modonna Center to co-design the study protocol (the content and delivery format of the exercise programs, recruitment and retention procedures and strategies, and procedures of study assessments).

The research team and the community advisory group (n=10) met weekly with the goal of making FE-SaLiR appealing to older Latino adults while maintaining the integrity of Chinese medicine exercises. Areas modified include the sequence of the exercises, difficulty level of the exercises, verbal instruction, background music, and visual aids (as compared to the official video published by the General Administration of Sport of China), etc. An English instruction video with the modified components was developed for phase 2 of the proposed study.

The group identified the barriers and enablers in health promotion programs for low-income, low-literacy, minority populations, and develop the strategies to engage and motivate the study participants.

The advisory group also guided the investigators in developing a process evaluation plan that provides insightful information on the acceptability of FE-SaLiR from the study participants in Phase 2 of the proposed study.

Phase 2: Pilot Intervention

Using a three-arm design, 3 senior centers were assigned to one of three conditions: 1) Wu Qin Xi and Ba Duan Jin unmodified; 2) FE-SaLiR: the modified Wu Qin Xi and Ba Duan Jin; 3) active control. The interventions will be delivered from February 2020 to May 2020. A total of 60 senior adults were expected to be enrolled in the study at baseline.

Data collection will be conducted at baseline and immediate post-intervention and include measures on physical and cognitive function, biometrics, health surveys, and mindfulness.

Recruitment: Participant recruitment started 1-month before the intervention by sending recruitment packets to senior centers. This packet includes a study information sheet, a recruitment flyer, and an informed consent form.

Process Evaluation: The process evaluation is informed by Phase I formative study. Qualitative and quantitative information on class attendance, home-exercise logs, class observation checklist, and participant's evaluation of the exercise will be collected. Focus group discussions will also be conducted regarding participants' experiences and with the goal of obtaining their input in planning a senior-friendly physical activity program.

ELIGIBILITY:
Inclusion Criteria:

* participating in Senior programs at Ella Austin, Good Samaritan, and Palacio del sol
* ages greater than 60
* ability to exercise in a standing position
* owning a cell phone or living with someone owning a cell phone
* willingness to complete a 3-month study

Exclusion Criteria:

* without permission to exercise from physicians
* inability to complete the 3-month study due to external factors

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-05-06 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Health-Related Quality of Life | Baseline and 12-week posttest
  The participants will complete SF-12 survey in self-administration or interview format. The SF-12 survey contains 12 items that focus on generic assessment on health-related quality of life.
Changes in Five-time Sit to Stand Test | Baseline and 12-week posttest
  The participants will to try stand up straight from the sitting position five times as quickly as they can for 5 times, without stopping between to assess their functional lower extremity strength, transitional movements, balance, and fall risk. Participants will be timed in seconds.

SECONDARY OUTCOMES:
Changes in Hand Grip Strength | Baseline and 12-week posttest
  The participant will hold the dynanometer in the hand and grip as hard as they can for twice for both hands, with a 10-20 seconds break between each trial. The average of number shown on the dynanometer indicates their grip strength (in kilogram) for each hand.
Changes in 6-minute Walking for Distance Test | Baseline and 12-week posttest
  Within 6 minutes, the participant will try to walk as far as possible. The distance (in meters) will be measured by a surveyor's wheel. Pre- and post-waling pain level and post-walking physical exertion level will be asked and recorded.
Changes in 50-feet Fast Walking Test | Baseline and 12-week posttest
  Two cones with a distance of 25 ft will be set and the participant will walk back and forth between the cones for a distance of 50 ft and try to walk as fast as possible without running. Time will be taken in seconds.
Changes in Lead Forward Balance Test | Baseline and 12-week posttest
  The participant will stand straight and reach forward. The moving distance of the finger tips will be measured in meters.
Changes in Resting Blood Pressure | Baseline and 12-week posttest
  The participant will sit in a chair with feet flat on the ground. After resting for 5 minutes, the blood pressure will be measured, repeated three times. The average systolic and diastolic blood pressure will be taken.
Changes in Height and Weight | Baseline and 12-week posttest
  Height and weight will be measured without clothes and shoes. Each participant will be measured for twice for both measures, height in meters and weight in kilograms, both to the nearest 0.1. If the difference for height measures were greater than 0.5 cm or the weight measures were greater than 0.25 kg, a third measure will be taken.
Changes in Pain Severity and Pain Functioning | Baseline and 12-week posttest
  The Brief Pain Inventory questionnaire will be provided in both English and Spanish, which contains 4 pain items and 7 interference items. The questionnaire will be conducted in an interview or self-administration format.
Changes in Mindfulness Skills | Baseline and 12-week posttest
  The 5-facet questionnaire, which contains 39 items can provide an estimate of mindfulness and self-awareness. The survey is completed through an interview for Spanish speakers. English speakers can complete the questionnaire either by self-administration or interview.
Changes in Symbol Digit Modalities Test | Baseline and 12-week posttest
  The participant will conduct the Symbol Digit Modalities Test to detect cognitive impairment. After being provided with instructions and a practice trial, the participant will complete the test in 90 seconds. Instructions will be orally presented in English or Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Zenong Yin, PhD, Principal Investigator — The University of Texas at San Antonio; Martha Martinez, MSN, RNC, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Yin Z, Martinez CE, Li S, Martinez M, Peng K, Land WM, Ullevig SL, Cantu A, Falk S, Hernandez AE, Ortega C, Parra-Medina D, Simmonds MJ. Adapting Chinese Qigong Mind-Body Exercise for Healthy Aging in Older Community-Dwelling Low-income Latino Adults: Pilot Feasibility Study. JMIR Aging. 2021 Nov 1;4(4):e29188. doi: 10.2196/29188. PMID 34723824